CLINICAL TRIAL: NCT04945135
Title: Controlled Donors After Circulatory Death and Brain Death: a Multicenter Study of
Brief Title: Controlled Donors After Circulatory Death and Brain Death: a Multicenter Study of Transfusion, One-year Graft Survival and Mortality. Cohort Study,
Status: Completed | Type: Observational
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Principal Investigator, Annabel Blasi, Consultor 1, Hospital Clinic of Barcelona
Other Study IDs: HCB/2019/1160
Record Dates: First submitted 2021-06-25; First posted 2021-06-30 (Actual); Last update posted 2021-06-30 (Actual); Status verified 2021-06

CONDITIONS: Liver Transplant

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- liver donors

SUMMARY:
RBC requirement ein DBD and DCD liver transplants

DETAILED DESCRIPTION:
Background: Controlled donation after cardiac circulatory death (cDCD) is accepted to expand the donor pool for liver transplantation (LT). However, transfusion requirements and perioperative outcomes should be elucidated. The aims of this multicentre study are to assess the red blood cell (RBC) transfusions, one-year graft and patient survival after LT with cDCD compared to donors after brain dead (DBD).

Methods: 591 LT patients conducted in ten centers during 2019 were reviewed. Thromboelastometry was used to manage coagulation and blood product transfusion in all centres. Normothermic regional perfusion was the standard technique for organ recovery.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing LT

Exclusion Criteria:

* acute liver failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients undergoing LT
Sampling Method: Non-Probability Sample
Enrollment: 591 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2021-06-25 (Actual)

PRIMARY OUTCOMES:
RBC transfusion | intraoperative

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Hospital de Cruces, Bilbao

IPD SHARING:
Plan to Share IPD: No